CLINICAL TRIAL: NCT05593588
Title: Senolytics as a Novel Treatment for Interstitial Lung Disease in Common Variable Immunodeficiency (CVID)
Brief Title: Senolytics Treatment of Interstitial Lung Disease in Common Variable Immunodeficiency
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Avni Joshi (Other)
Responsible Party: Sponsor-Investigator, Avni Joshi, Regulatory Sponsor and Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-003119
Record Dates: First submitted 2022-10-21; First posted 2022-10-25 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Common Variable Immunodeficiency; Interstitial Lung Disease Due to Systemic Disease
MeSH Terms: conditions — Common Variable Immunodeficiency | interventions — fisetin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fisetin Group (Experimental): Subjects will receive the supplement, Fisetin, for 2 cycles of 2 consecutive days (first on days 0 & 1 and then repeated on days 28 & 29)
  Interventions: Drug: Fisetin
- Placebo Group (Placebo Comparator): Subjects will receive placebo for 2 cycles of 2 consecutive days (first on days 0 & 1 and then repeated on days 28 & 29)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fisetin — 20 mg per kilogram (kg) of body weight supplied in 100 mg capsules and administered orally on days 0, 1, 28, and 29
  Arms: Fisetin Group
Drug: Placebo — Looks exactly like the study drug, but it contains no active ingredient. Administered orally on days 0, 1, 28 and 29
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to determine if the supplement, Fisetin, can be used as a treatment option for common variable immunodeficiency (CVID) by comparing its efficacy to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have received a diagnosis of CVID according to the international consensus document (ICON) at least 30 days before enrollment.
* Physician diagnosis of possible GLILD associated with CVID.
* IgA results.
* Female patient is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile. (A negative pregnancy test for women whose menopausal status is determined by self-reported absence of menstrual periods in the past 12 months will be required within 72 hours prior to randomization).
* Patient must be able and willing to comply with the requirements of this study protocol.

Exclusion Criteria:

* Unable or unwilling to give informed consent.
* Presence of any condition that the Investigator or the subject's attending physician believes would put the subject at risk or would preclude the patient from successfully completing the trial.
* Pregnant and/or lactating. Women of childbearing potential (WCBP) must have a negative pregnancy test within 72 hours prior to randomization.

WCBP who are unwilling to abstain from sex or use an adequate method of contraception from the time of the first IP administration through 48 hours after the last IP administration.

* Men who are unwilling to abstain from sex with WCBP or use an adequate method of contraception from the time of the first IP administration through 48 hours after the last IP administration.
* Prisoners, institutionalized individuals, or others who may be considered vulnerable populations, such as individuals with dementia.
* Patient currently hospitalized or under immediate consideration for hospitalization.
* Current use of tobacco products or as per clinical judgement.
* Current excessive caffeine intake (400 mg or more per day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in immunophenotyping of peripheral T lymphocytes | Baseline, 6 months
  Measured by percentage of activated CD4+25+ T cells

SECONDARY OUTCOMES:
Change in Forced Vital Capacity (FVC) | Baseline, 6 months
  Measured by spirometry to determine the maximal amount of air that can be forcibly exhaled from the lungs after a full inhale, reported as liters (L)
Change in radiologic imaging in subjects | Baseline, 3 months, 6 months
  Number of subjects to have a 10% improvement with the CT scoring system. Radiologist will score the CT scans at each time point and changes in score at each time point will be noted.
Use of MRI imaging for assessment of GLILD | 6 months
  Number of MRI images that were used to assess for GLILD compared to High-resolution Computed Tomography (HRCT) use
Infectious complications | 6 months
  Number of subjects to experience infectious complications
Adverse Events | 6 months
  Number of adverse events reported
Change in quality of life | Baseline, 6 months
  Measured using the RAND 36-Short Form Survey Instrument (SF-36). The SF-36 Health Survey is a 36-item, participant-reported survey that measures patient health and disability. Possible scores range from 0 to 100, with 0 indicating maximum disability, and 100 indicating no disability
Change in 6 minute walk test | Baseline, 6 months
  Number of subjects to have a 10% improvement in 6 minute walk test. The 6 minute walk test measures the distance a person is able to walk in 6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Avni Joshi, MD, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials